CLINICAL TRIAL: NCT02855580
Title: Integrating Pharmacogenomic Testing Into a Child Psychiatry Clinic
Acronym: PGX
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201601035
Record Dates: First submitted 2016-07-19; First posted 2016-08-04 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Obsessive Compulsive Disorder; Major Depressive Disorder; Anxiety
Keywords: Pharmacogenomic; child; psychiatry; Obsessive Compulsive Disorder; Depression; Anxiety; CYP2D6; CYP2C19; Selective serotonin reuptake inhibitor; SSRI
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Depressive Disorder, Major; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PGX Testing Based Treatment: Treatment will be administered based on the results that are obtained from the pharmacogenomics testing. Results from testing will be provided two weeks after specimen collection.
- Standard of Care Treatment: Treatment will be based off of the standard of care. Results from pharmacogenomics testing will be provided at the end of the study.

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability, and utility of pharmacogenomic (PGX) testing (specifically for the cytochrome P450 2D6 and 2C19 genes) prior to initiating treatment with an antidepressant (AD) among children and adolescents in the University of Florida Child Psychiatry clinics.

DETAILED DESCRIPTION:
This project will assess the feasibility of implementing pharmacogenomic testing (PGX) for specific genes involved in the metabolism of antidepressants (CYP2D6 and CYP2C19) into the child psychiatry clinic at UF.

Although not widely implemented to date, naturalistic studies in adult psychiatry populations have shown that PGX testing can improve patient outcomes, increase medication adherence, and reduce costs. However, there have been no studies of psychiatry-focused PGX testing in children. One in every four children and adolescents suffers from a mental illness (more than half have a mood or anxiety disorder) that is severe enough to impact their functioning at school, at home, or in other important areas. Although psychotherapy remains the first line treatment for children with mild or uncomplicated symptoms, the use of psychotropic medications in children has increased steadily over the last decade. These medications are effective for many children, but carry a substantial risk of side effects, including gastrointestinal, cognitive, systemic, and psychiatric (including treatment emergent suicidal ideation). For most treatment responders, improvement is typically seen four to eight weeks after the target dose has been achieved (twelve weeks for obsessive compulsive disorder). Thus, identifying the best medication options prior to treatment initiation could decrease the likelihood of side effects severe enough to require medication discontinuation or changes, and minimize the time to response. In this study, 50 children and adolescents with major depression, anxiety, or obsessive compulsive disorders who are beginning treatment with a new antidepressant will be recruited and PGX testing will be conducted. Twenty five children will be randomized to receive PGX testing prior to starting/changing medications and 25 to receive treatment as usual (these children will receive their PGX results at the end of 12 weeks). Members of the UF Health Personalized Medicine Program will provide education to the prescribing clinicians about PGX testing and will create patient-specific consultations regarding the PGX results.

Assess clinicians' and parents' willingness to use PGX testing in making treatment decisions, as well as their knowledge and beliefs about PGX testing (pre-and post-study). Also assess, as pilot data for a larger randomized controlled trial, differences in side effect profiles, treatment adherence, and symptom improvements between the PGX cases and controls.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 8 to 20 years old
* Have been diagnosed with and receiving treatment for mood disorder, anxiety, or obsessive compulsive disorder
* Receiving treatment at UF child psychiatry clinic

Exclusion Criteria:

* Children with a primary diagnosis of autism
* High risk for suicide
* Children determined by UF psychiatrist to be too ill to tolerate waiting two weeks to begin medication treatment

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consists children and adolescents ages 8 to 20 who are receiving medication treatment for a mood disorder, anxiety disorder, or obsessive compulsive disorder.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Antidepressant Tolerance | From week 0 through week 12
  The feasibility of pharmacogenomic (PGX) testing (specifically for the cytochrome P450 and 2C19 genes) prior to initiating treatment in a child and adolescent population will be measured through medication compliance and frequency of medication changes as described in the patient's medical record.

SECONDARY OUTCOMES:
Symptom Severity-Depression | From week 0 through week 12
  Depression will be assessed using the Children's Depression Inventory (CDI)
Symptom Severity-Anxiety | From week 0 through week 12
  Anxiety will be assessed using the Screen for Child Anxiety Related Emotional Disorders (SCARED)
Symptom Severity-Obsessive Compulsive Symptoms | From week 0 through week 12
  Obsessive compulsive symptoms will be assessed using the Children's Florida Obsessive Compulsive Inventory (C-FOCI).
Side effects | From week 1 through week 12
  Assess effects associated with AD treatment using a standardized questionnaire commonly used in clinical trials of children and modified for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mathews, MD, Principal Investigator — University of Florida
Locations (1):
- Child Psychiatry Clinic at University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Carol A. Mathews, MD Research Lab Information — http://pgenes.net/